CLINICAL TRIAL: NCT06226961
Title: Immediate Effects of Dynamic Cupping on Shoulder Active Range of Motion of Senior Male Handball Athletes: A Randomized Controlled Trial
Brief Title: Effects of Dynamic Cupping on Shoulder Active Range of Motion of Senior Male Handball Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FISIO-3-29072019
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-01

CONDITIONS: Healthy
MeSH Terms: interventions — Cupping Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): For the dynamic cupping protocol, the participants will be instructed to remain seated on the massage table with their feet supported, and the technique will applied to the entire shoulder (anterior, lateral and posterior face) and surrounding muscles (upper trapezius and pectoralis major). The cupping will be performed using a plastic cupping cup (5,08 cm in diameter) (K.S. Choi Corp®) and a pistol grip hand pump (K.S. Choi Corp®). The dynamic cupping will be performed for ten minutes, at a slow pace, and consists of applying a small amount of massage cream (ATL®) over the entire shoulder (to obtain the ideal sliding surface for cupping application), insufflation of the suction cup, with two pumps, and sliding it in the direction of the muscle fibers around the shoulder and also in the transversal direction.
  Interventions: Device: cupping
- Control group (No Intervention): Participants in the CG group will remain at rest, sitting on the massage table for 10 minutes.

INTERVENTIONS:
Device: cupping — The dynamic cupping will be performed for ten minutes, at a slow pace, and consisted of applying a small amount of massage cream (ATL®) over the entire shoulder (to obtain the ideal sliding surface for cupping application), insufflation of the suction cup, with two pumps, and sliding it in the direction of the muscle fibers around the shoulder and also in the transversal direction.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to to verify the immediate effects of dynamic cupping on shoulder active range of motion (AROM) of senior male handball athletes.

DETAILED DESCRIPTION:
After completing the questionnaire, 80 senior male handball athletes will be randomly divided into two designated groups, Intervention Group (IG; n = 40) (dynamic cupping therapy) and Control Group (CG; n = 40) (no intervention).

Shoulder AROM (flexion, extension, abduction, adduction, horizontal adduction, horizontal abduction, internal rotation and external rotation movements) will be assessed in both control and intervention groups before (M0) and after (M1) intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy senior handball athletes in competition with at least three training sessions per week.

Exclusion Criteria:

* history of injury, fracture or surgical intervention in the upper limb in the last six months before the study;
* vestibular, neurological or cardiorespiratory diseases;
* reported pain in the upper limb or spine
* presence of contraindication for cupping (deep venous thrombosis, with active infection or open wound.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
active movements of the shoulder | [Time Frame: Change from Baseline (M0) to Immediately after intervention or control (M1)]
  Data will be collected in two moments: baseline (M0) and after the intervention/control (M1). The shoulder range of motion will be measured using a universal goniometer.
  Participants will be instructed to perform the various active movements of the shoulder on the dominant upper limb. The assessments of the shoulder flexion, extension, abduction and adduction movements will be performed standing up, controlling possible compensations. To assess abduction and horizontal adduction movements, the participants will remain seated on a massage table. Internal and external rotation movements will be assessed on a massage table in supine, without inclination. Measurements will be considered invalid if the participant is compensated with another body part. Three measures will be collected for each movement and the average of the three will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior Saúde Fernando Pessoa, Porto, Portugal